CLINICAL TRIAL: NCT02313389
Title: Phase III Trial Evaluating Maintenance Treatment Versus Observation in Elderly Patients Suffering From Primary Central Nervous System Lymphoma in Complete Remission After High Dose Methotrexate Based Chemotherapy in First Line
Brief Title: Maintenance Treatment Versus Observation in Elderly Patients With PCNS Lymphoma
Acronym: BLOCAGE-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130950; 2014-002597-37 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — Rituximab; Methotrexate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- maintenance chemotherapy (Experimental): Clinical examination and MRI will be performed every 3 months for 2 years and then every 6 months until tumor progression.
  Neurocognitive tests will be performed at randomization and annually. Quality of life questionnaires at randomisation and every 3 months
  Interventions: Drug: Rituximab, Methotrexate, Temozolomide
- observation (No Intervention): Clinical examination and MRI will be performed every 3 months for 2 years and then every 6 months until tumor progression.
  Neurocognitive tests will be performed at randomization and annually. Quality of life questionnaires at randomisation and every 3 months

INTERVENTIONS:
Drug: Rituximab, Methotrexate, Temozolomide — Seven monthly R-MT cycles including high dose MTX (3.5g/m2, D1), TMZ, rituximab.
  Arms: maintenance chemotherapy

SUMMARY:
Hypothesis

Our hypothesis is that maintenance chemotherapy will prolong complete remission obtained after a standard induction chemotherapy with an acceptable toxicity in the elderly.

Rationale

* Treatment of the elderly is challenging, indeed age over 60 is associated both with a poor prognosis and a high risk of treatment induced neurotoxicity with devastating consequences on quality of life. Therefore it has become standard practice to treat elderly in first line with high-dose methotrexate (MTX) based polychemotherapy alone, avoiding whole brain radiotherapy (WBRT) or deferring it for recurrence.
* There is a clear need to improve disease control after induction chemotherapy. Since consolidation with WBRT or intensive chemotherapy with autologous stem cell rescue are either poorly effective and/or too toxic in the elderly population, maintenance chemotherapy is an interesting alternative approach. Several agents, such as high-dose MTX, temozolomide (TMZ), rituximab, with a reported activity in PCNSL and acceptable safety profile, as single agent or combined, are good candidates for maintenance

DETAILED DESCRIPTION:
Objectives

* The primary objective is to evaluate the benefit estimated by the PFS associated with maintenance chemotherapy compared to observation in patients ≥ 60 years having achieved a complete response after a high-dose MTX based induction chemotherapy
* The secondary objectives are to assess:

  * Overall survival
  * Safety of maintenance chemotherapy
  * Neurocognitive outcome
  * Quality of life of the patients

Inclusion and exclusion criteria

At registration

* Inclusion criteria

  * Newly diagnosed primary cerebral lymphoma
  * Age >60 years
  * Pathology proven diagnosis
  * Positive cytology of the CSF or vitreous
  * Karnofsky Performance Status >40
  * No evidence of systemic NHL (body CT scan, bone marrow biopsy)
  * Adequate haematological, renal and hepatic function
  * Calculated creatinine clearance > 40 ml/min
* Non inclusion criteria

  * Positive HIV serology
  * Preexisting immunodeficiency (organ transplant recipient)
  * Prior treatment for PCNSL
  * Isolated primary intra-ocular lymphoma
  * Low grade lymphoma
  * Any other active primary malignancy

At randomization

* Complete response on MRI after induction chemotherapy according to the IPCG criteria
* Karnofsky Performance Status >40
* Adequate haematological, renal and hepatic function

Study Design

* This study is an open label multicenter randomized phase III trial comparing maintenance chemotherapy versus observation in complete responders to high dose MTX based induction chemotherapy.
* Patients are registered to participate in the study at time of initial diagnosis and study enrolment before the induction chemotherapy.
* Induction chemotherapy (R-MPVA protocol) includes 4 to 5 monthly cycles of high dose MTX (3.5g/m2, D1 and D15), procarbazine, vincristine, rituximab followed by one cycle of high dose cytarabine consolidation.
* Randomization to observation (arm 1) or maintenance (arm 2) will be carried out only for patients in complete response (CR) after induction chemotherapy Arm 1: Observation Arm 2: Seven monthly R-MT cycles including high dose MTX (3.5g/m2, D1), TMZ, rituximab

Sample size, duration of the study, feasibility

* 295 patients need to be enrolled to randomize 192 patients
* Duration of the study: 6 years (accrual period= 4 years; minimal follow-up = 2 years)

  26 participating expert centers from the national LOC network

The trial is supported by the neurooncology ANOCEF and the lymphoma LYSA clinical research groups.

Ancillary study LOCALYSE:

Role of [18F]-FDG brain PET in newly diagnosed primary cerebral lymphoma, in immunocompetent patient older than 60 years

Rationale Patients older than 60 years account for half of cases of PCNSL and have a poorer outcome. No prognostic or predictive factors exist for survival after initial remission. [18F]FDG-PET (Fluoro Deoxy Glucose) plays a key role in grading and therapy monitoring of systemic diffuse large B-cell type.

LOCALYZE is an ancillary PET/MR clinical study from BLOCAGE 01. The aim is to evaluate the usefulness of [18F]FDG-PET to monitor treatment response in PCNSL (Primary Central Nervous System Lymphoma) older than 60 years (n=56), in complement to multiparametric MRI.

Hypothesis We assume that the development of new imaging biomarker extracted from PET imaging and multiparametric MRI, could improve the assessment of treatment response in PCNSL.

Primary aim To evaluate the predictive value of [18F]FDG-PET assessment performed at the end-of-treatment (high-dose methotrexate based polychemotherapy), on progression free survival in newly diagnosed PCNSL with age ≥60 years (n=56).

Primary Outcome Measures:

Progression free survival calculated from the date of completion of the end of chemotherapy PET

Study design

Three [18F]-FDG PET/MR will be performed in the Department of Nuclear Medicine - Pitié-Salpêtrière Hospital:

* prior to initiation of R-MPVA chemotherapy (Rituximab Methotrexate Procarbazine Vincristine Aracytine ) (PET#1),
* after two chemotherapy cycles (PET#2),
* at the end of the first-line chemotherapy regimens (PET#3).

Inclusion criteria (=Blocage-01) Blocage01 eligibility

Exclusion criteria

* Uncontrolled diabetes with fasting glycaemia > 200 mg/dL
* Sensitivity to active substance in [18F]-FDG
* Calculated creatinine clearance < 40 ml/min
* No contraindication to MRI

ELIGIBILITY:
Inclusion criteria At registration Inclusion criteria

* newly diagnosed primary cerebral lymphoma
* Age ≥60 years
* Pathology proven diagnosis or positive cytology of the CSF or vitreous
* Karnofsky Performance Status ≥40
* No evidence of systemic NHL (body CT scan, bone marrow biopsy)
* Adequate haematological, renal and hepatic function
* Calculated creatinine clearance > 40 ml/min

At randomization

* Complete response on MRI after induction chemotherapy according to the IPCG criteria
* Karnofsky Performance Status ≥40
* Adequate haematological, renal and hepatic function

Exclusion criteria

* Positive HIV serology
* Preexisting immunodeficiency (organ transplant recipient)
* Prior treatment for PCNSL
* Isolated primary intra-ocular lymphoma
* Low grade lymphoma
* Any other active primary malignancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2015-09; Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 6 years

SECONDARY OUTCOMES:
overall survival | 6 years
Toxicity graded according to the NCI-CTCAE | 6 years
  Toxicity graded according to the NCI-CTCAE
Cognitive functions evaluated by a standardized and validated test battery exploring 5 cognitive domains | 6 years
  Cognitive functions evaluated by a standardized and validated test battery exploring 5 cognitive domains
Quality of life | 6 years
  Quality of life assessed by the EORTC QLC-C30 questionnaire and the brain cancer module (BCM20)

CONTACTS AND LOCATIONS:
Overall Officials: Khe HOANG-XUAN, Md, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitie Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rozenblum L, Houillier C, Baptiste A, Soussain C, Edeline V, Naggara P, Soret M, Causse-Lemercier V, Willems L, Choquet S, Ursu R, Galanaud D, Belin L, Hoang-Xuan K, Kas A. Interim FDG-PET improves treatment failure prediction in primary central nervous system lymphoma: An LOC network prospective multicentric study. Neuro Oncol. 2024 Jul 5;26(7):1292-1301. doi: 10.1093/neuonc/noae029. PMID 38366824